CLINICAL TRIAL: NCT07328230
Title: A Prospective Randomized Controlled Trial for Treatment of Idiopathic Hyperaldosteronism: Superselective Adrenal Arterial Embolization Versus Oral Spironolactone
Brief Title: Superselective Adrenal Arterial Embolization Versus Oral Spironolactone for Treatment of Idiopathic Hyperaldosteronism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Collaborators: Second Affiliated Hospital of Nanchang University (Other); First Affiliated Hospital of Chengdu Medical College (Other)
Responsible Party: Principal Investigator, Xiongjing Jiang, professor, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-1714
Record Dates: First submitted 2025-12-26; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Idiopathic Hyperaldosteronism; Hyperaldosteronism
Keywords: Superselective adrenal arterial embolization; Spironolactone; Hyperaldosteronism; Hypertension; Mineralocorticoid receptor antagonists(
MeSH Terms: conditions — Hyperaldosteronism; Hypertension | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Superselective Adrenal Arterial Embolization (Experimental): Patients in the experimental group will undergo percutaneous superselective adrenal arterial embolization.
  Interventions: Procedure: Superselective Adrenal Arterial Embolization
- Spironolactone (Active Comparator): Patients in this group will receive oral spironolactone.
  Interventions: Drug: Spironolactone

INTERVENTIONS:
Procedure: Superselective Adrenal Arterial Embolization — Patients in this group will undergo percutaneous superselective adrenal artery embolization (SAAE). Under fluoroscopic guidance, a microcatheter or an over-the-wire balloon catheter will be navigated into the target adrenal arteries, followed by the slow, controlled infusion of absolute ethanol to achieve localized tissue ablation.
  Arms: Superselective Adrenal Arterial Embolization
Drug: Spironolactone — Patients will be treated with spironolactone.
  Arms: Spironolactone

SUMMARY:
Idiopathic hyperaldosteronism (IHA) represents about 65% of primary hyperaldosteronism cases. Although mineralocorticoid receptor antagonists (MRAs) are the standard first-line treatment, they are often limited by adverse effects. Superselective adrenal artery embolization (SAAE) has been utilized for IHA over the last decade, yet comparative studies against MRAs are lacking. The objective of this study is to compare the safety and efficacy of SAAE and MRA to determine the feasibility of SAAE in treating IHA.

DETAILED DESCRIPTION:
Idiopathic hyperaldosteronism (IHA), characterized by bilateral adrenal hyperplasia, constitutes approximately 65% of primary hyperaldosteronism cases. While Mineralocorticoid Receptor Antagonists (MRAs) like spironolactone are the gold-standard medical therapy, their long-term use is frequently hampered by dose-dependent side effects, including gynecomastia, electrolyte imbalances, and renal insufficiency, leading to poor patient compliance.This study investigates Superselective Adrenal Artery Embolization (SAAE) as a minimally invasive interventional alternative. Unlike total adrenalectomy, SAAE targets specific terminal branches of the adrenal arteries to reduce aldosterone overproduction while preserving sufficient cortical function. Despite its clinical application over the last decade, high-quality comparative data between SAAE and pharmacological MRA therapy remain scarce.The primary objective of this research is to evaluate the safety and clinical efficacy of SAAE versus MRA through a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Aged from 15 to 60 with no limits in sex;
2. Patients are diagnosed with primary aldosteronism according to the criteria of the 2016 Endocrine Society guidelines;
3. Sub-typing diagnosis confirmed idiopathic hyperaldosteronism;
4. Patients or their legal representatives have to sign written informed consent approved by the ethics committee.

Exclusion Criteria:

1. Unilateral adrenal hyperplasia;
2. Renal insufficiency with an estimated glomerular filtration rate (based on the modification of diet in renal disease criteria) <45 ml/min/1.73 m², and/or serum creatinine >176 μmol/L；
3. Hemorrhagic or ischemic stroke, endovascular stent implantation and myocardial infarction within the previous 3 months;
4. Severe contrast agent allergy;
5. Women who are pregnant or planning to become pregnant;
6. Patients with other serious organic diseases cannot tolerate SAAE treatment;
7. Other forms of secondary hypertension.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 172 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of 24-h mean systolic blood pressure at 6 months compared with baseline. | 6 months after randomization
  change of 24-h mean systolic blood pressure at 6 months compared with baseline.

SECONDARY OUTCOMES:
Change of 24-h mean diastolic blood pressure at 6 months compared with baseline. | 6 months after randomization
  change of 24-h mean diastolic blood pressure at 6 months compared with baseline.
Change of office systolic and diastolic blood pressure at 1, 3, 6 months, 24-h mean systolic and diastolic blood pressure at 1, 3 months, compared with baseline | 1, 3, 6 months after randomization
  Change of office blood pressure at 1, 3, 6 months compared with baseline
change of antihypertensive medication burden at 1, 3, 6 months compared with baseline | 1, 3, 6 months after randomization
  change of antihypertensive medication burden at 6 months compared with baseline
Incidence of clinical events | 6 months after randomization
  Incidence of clinical events including: major adverse cardiovascular events(MACE), renal insufficiency, adrenal insufficiency, hyperkalemia, vascular complication, flank/back pain, gynecomastia, breast tenderness, sexual dysfunction,etc.
Change of Serum potassium at 3, 6 months after randomization, compared with baseline | 3,6 months after randomization
  Change of Serum potassium at 3, 6 months compared with baseline
Change of plasma aldostrone, renin, cortisol concentration at 3, 6 months compared with baseline | 3, 6 months after randomization
  Change of plasma aldostrone, renin, cortisol concentration at 3, 6 months compared with baseline
Change of estimated glomerular filtration rate(eGFR) and at 3, 6 months compared with baseline | 3, 6 months after randomization
  Change of estimated glomerular filtration rate(eGFR) and at 3, 6 months compared with baseline

CONTACTS AND LOCATIONS:
Overall Officials: Xiongjing Jiang, MD, Principal Investigator — Fuwai Hospital, National Center for Cardiovascular Disease
Locations (3):
- China (3):
  - Fuwai Hospital, National Center for Cardiovascular Disease, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality
  - Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Affiliated Hospital of Chengdu Medical College, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dong H, Zou Y, He J, Deng Y, Chen Y, Song L, Xu B, Gao R, Jiang X. Superselective adrenal arterial embolization for idiopathic hyperaldosteronism: 12-month results from a proof-of-principle trial. Catheter Cardiovasc Interv. 2021 May 1;97 Suppl 2:976-981. doi: 10.1002/ccd.29554. Epub 2021 Feb 19. PMID 33605538
- [Result] Zhao Z, Liu X, Zhang H, Li Q, He H, Yan Z, Sun F, Li Y, Zhou X, Bu X, Wu H, Shen R, Zheng H, Yang G, Zhu Z; Chongqing Endocrine Hypertension Collaborative Team. Catheter-Based Adrenal Ablation Remits Primary Aldosteronism: A Randomized Medication-Controlled Trial. Circulation. 2021 Aug 17;144(7):580-582. doi: 10.1161/CIRCULATIONAHA.121.054318. Epub 2021 Aug 16. No abstract available. PMID 34398686